CLINICAL TRIAL: NCT00614133
Title: Hypocaloric Isonitrogenous Nutrition and Epidural Analgesia: a Novel Strategy to Induce Anabolism After Surgery
Brief Title: Effect of Intravenous Nutrition and Epidural Analgesia on Protein Loss After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Thomas Schricker, Department of Anaesthesia, Royal Victoria Hospital, MUHC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MOP-64456
Record Dates: First submitted 2008-01-30; First posted 2008-02-13 (Estimated); Last update posted 2008-02-13 (Estimated); Status verified 2008-01

CONDITIONS: Postoperative Protein Catabolism
Keywords: protein metabolism; surgery; parenteral nutrition
MeSH Terms: conditions — Hyperphagia | interventions — Glucose; Amino Acids

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Preoperative nutrition.
  Interventions: Other: Intravenous nutrition with glucose and amino acids
- 2 (Active Comparator): Preoperative fasting.
  Interventions: Other: Intravenous nutrition with glucose and amino acids.

INTERVENTIONS:
Other: Intravenous nutrition with glucose and amino acids — Glucose and amino acids intravenously starting 20 hours before the operation until the second postoperative day. Glucose provides 50% and amino acids 20% of each patient's measured resting energy expenditure.
  Arms: 1
Other: Intravenous nutrition with glucose and amino acids. — Glucose and amino acids intravenously starting with surgical skin incision until the second postoperative day. Glucose provides 50% and amino acids 20% of each patient's measured resting energy expenditure.
  Arms: 2

SUMMARY:
Loss of muscle mass and body protein are the main causes of fatigue after bowel surgery, which may result in a longer hospital stay and a higher rate of complications. This particularly applies to malnourished patients with cancer who undergo surgery with less muscle protein reserves than patients who are well-nourished. Anesthesiologists can favourably influence these undesirable consequences of surgery by choosing the type of pain treatment, i.e. analgesia. Our group recently observed that pain treatment with epidural catheters (these are placed in the so called epidural space, which lies between the spine and the skin of the back), in contrast to the more conventional use of intravenous morphine, can prevent the loss of body protein after surgery.

The goal of the present research program is to study whether this protein sparing effect of epidural analgesia can be further augmented if we feed our patients intravenously with glucose and protein starting the day prior to surgery. We believe that this new concept will not only avoid the increased protein loss after surgery, but will also help patients to build up new protein which is needed to fight the stress caused by the operation.

DETAILED DESCRIPTION:
The major objective of the nutritional management of surgical patients is to accelerate wound healing and increase resistance to infection while preventing wastage of functional and structural proteins. Parenteral nutrition represents a useful strategy to achieve this goal, particularly in patients undergoing major abdominal procedures with temporary intolerance to oral feeding. At present administration of large, hypercaloric amounts of glucose together with amino acids is the only nutritional modality to establish a positive protein balance (anabolism) after surgery. The fact that hyperalimentation requires central venous cannulation, causes hyperglycemia and is associated with increased morbidity is an impediment to its routine use. Attempts to induce anabolism by diminishing the glucose load to iso- or hypocaloric quantities failed because of

* failure to control for type and quality of perioperative analgesia
* inadequate assessment of the patient's catabolic status prior to surgery with subsequent
* lack of individualization of energy and substrate supply.

We recently demonstrated that segmental pain relief by epidural analgesia facilitates oxidative glucose utilization thereby decreasing the amount of glucose necessary to attenuate protein losses after surgery. Hypocaloric glucose and epidural analgesia prevented the postoperative increase in protein oxidation, but only if preoperative fasting was avoided, i.e. the glucose infusion was started 24 hours before surgery. We also showed that patients with epidural analgesia could be rendered anabolic by short term administration of glucose and amino acids. Based on our findings of anti-catabolic and anabolic effects of epidural analgesia in the presence of energy and substrate supply we now propose that epidural analgesia and hypocaloric parenteral nutrition initiated 24 hours before colorectal surgery will produce a more positive postoperative protein balance including a greater muscle protein synthesis than when initiated with skin incision.

In order to test the validity of this assumption, patients scheduled for elective colorectal cancer surgery will be randomly assigned to an "early" or "late" feeding protocol. "Early" nutrition will start 24 hours prior to surgery, "late" nutrition will commence with surgical skin incision. Nutrition will be adjusted to provide 50% of the patient's actual energy expenditure as glucose and 20% as amino acids. The stable isotope tracer L-[1-13C]leucine will be applied to assess whole body protein breakdown, amino acid oxidation and protein synthesis. A positive protein balance (difference between protein synthesis and protein breakdown) will be used as an indicator of anabolism. Because whole body protein kinetics provide no insight into metabolic processes at organ level (muscle, liver), the fractional synthesis rates of albumin, fibrinogen and muscle protein will also be determined after surgery.

The demonstration of anabolic effects of epidural analgesia and nutrition with less than half the commonly used energy would have a valuable practical application. If the nutrient load can be decreased, use can be made of peripheral veins and hyperglycemia can be avoided, thus making nutritional therapy more efficacious, safer and available to more patients.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists <3
* colorectal surgery for non-metastatic colorectal carcinoma including right and left hemicolectomy, transverse, subtotal and total colectomy, sigmoid resection
* ability to give informed consent

Exclusion Criteria:

* signs of severe malnutrition or obesity: body mass index <18 or >25 >10% involuntary body weight loss over the preceding 6 months serum albumin <21 g/L
* significant cardiorespiratory, hepatic, renal and neurological disease
* ingestion of drugs known to affect protein, glucose and lipid metabolism (for example steroids)
* musculoskeletal or neuromuscular disease
* severe anemia (hemoglobin <10 g/dL)
* pregnancy
* history of severe sciatica or back surgery or other conditions which contraindicate the use of epidural catheters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2004-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
protein balance | two days after surgery

SECONDARY OUTCOMES:
albumin synthesis, fibrinogen synthesis, total plasma protein synthesis, mRNA expression of ubiquitin | two days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P Schricker, MD PhD, Principal Investigator — Department of Anaesthesia, McGill University Health Centre
Locations (1):
- Royal Victoria Hospital, McGill University Health Centre, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Schricker T, Meterissian S, Lattermann R, Adegoke OA, Marliss EB, Mazza L, Eberhart L, Carli F, Nitschman E, Wykes L. Anticatabolic effects of avoiding preoperative fasting by intravenous hypocaloric nutrition: a randomized clinical trial. Ann Surg. 2008 Dec;248(6):1051-9. doi: 10.1097/SLA.0b013e31818842d8. PMID 19092350